CLINICAL TRIAL: NCT07307547
Title: A Multi-center, Randomized, Controlled Clinical Study on the Efficacy of Artificial Intelligence-Assisted Colonoscopy in Improving the Screening of Colorectal Cancer and Precancerous Lesions.
Brief Title: Efficacy of AI-Assisted Colonoscopy for Screening Colorectal Neoplasia (AI-COLOSCREEN)
Acronym: AI-COLOSCREEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Clinical professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2025-0756
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Neoplasms; Colonic Polyp; Adenoma; Colorectal Cancer
Keywords: Artificial Intelligence; Colonoscopy; Colorectal Cancer Screening; Adenoma Detection Rate; Deep Learning
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: AI-Assisted Colonoscopy (Experimental): Participants will undergo a high-definition colonoscopy procedure where a real-time artificial intelligence system analyzes the video feed to assist the endoscopist in identifying and highlighting suspicious lesions.
  Interventions: Device: AI-Assisted Colonoscopy
- Control: Conventional Colonoscopy (No Intervention): Participants will undergo a standard high-definition colonoscopy procedure performed by a qualified endoscopist without the assistance of the artificial intelligence system. The AI software will not be active during these procedures.

INTERVENTIONS:
Device: AI-Assisted Colonoscopy — High-definition colonoscopy procedure with a real-time video analyzed artificial intelligence system.
  Arms: Experimental: AI-Assisted Colonoscopy

SUMMARY:
This study is a multi-center, randomized controlled trial designed to evaluate whether an artificial intelligence (AI) system can assist endoscopists to improve the detection rate of colorectal adenomas and cancers during colonoscopy compared to standard colonoscopy. Early screening and diagnosis are key to reducing the burden of colorectal cancer, but current colonoscopy has limitations, including the risk of missed lesions. This trial aims to determine if AI can enhance screening quality and diagnostic accuracy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening is crucial for early detection and reducing mortality, yet current colonoscopy techniques face challenges such as variable adenoma detection rates (ADR) and the risk of missed diagnoses for subtle lesions. This study is a prospective, multi-center, parallel-group, randomized controlled trial aiming to validate the clinical value of an AI-assisted diagnostic system in improving screening quality. A total of 3342 participants will be randomized in a 1:1 ratio to undergo either AI-assisted colonoscopy (Experimental Group) or conventional high-definition colonoscopy (Control Group). The primary objective is to compare the ADR between the two groups. Secondary objectives include assessing the detection rate of advanced or specific types of polyps, the mean number of adenomas per procedure, and the impact of the AI system on both patient and physician satisfaction. The study will provide high-quality evidence for the standardized application of AI technology in CRC screening, with the ultimate goal of reducing the incidence and mortality of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive.
2. Scheduled for a screening, diagnostic, or surveillance colonoscopy.
3. Able to understand the study protocol and provide written informed consent.

Exclusion Criteria:

1. Known contraindications to colonoscopy or biopsy.
2. Personal history of colorectal cancer, inflammatory bowel disease (IBD), or previous colorectal surgery.
3. Known or suspected colorectal polyposis syndrome (e.g., Familial Adenomatous Polyposis - FAP).
4. Patients with active colorectal bleeding, bowel obstruction, or toxic megacolon.
5. Women who are pregnant, planning to become pregnant, or are breastfeeding.
6. Participation in another interventional clinical trial within the 30 days prior to enrollment.
7. Any other condition that, in the investigator's judgment, would make the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3342 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | From the day of the procedure up to 14 days post-procedure.
  The proportion of participants with at least one histologically confirmed colorectal adenoma or adenocarcinoma. Detection and specimen collection occur during the colonoscopy, with final confirmation based on pathology reports.

SECONDARY OUTCOMES:
Mean Adenomas Per Colonoscopy (APC) | From the day of the procedure up to 14 days post-procedure.
  The mean number of histologically confirmed adenomas detected per participant. The number of polyps is counted during the procedure, but confirmation of adenoma status depends on pathology.
Advanced Adenoma and Sessile Serrated Adenoma/Polyp (SSA/P) Detection Rate | From the day of the procedure up to 14 days post-procedure.
  The proportion of participants with at least one histologically confirmed advanced adenoma (defined as ≥10mm, or with high-grade dysplasia or villous components) or SSA/P.
Patient Satisfaction Score | Assessed within 1 hour after completion of the colonoscopy procedure.
  Assessed using a 5-point Likert scale questionnaire evaluating examination comfort and acceptance of the AI system (1=very unsatisfied, 5=very satisfied).
Physician Satisfaction Score | Assessed within 1 hour after completion of the colonoscopy procedure.
  Assessed using a 5-point Likert scale questionnaire evaluating the AI system's usability and reliability (1=very unsatisfied, 5=very satisfied).
Incidence of Procedure-Related Adverse Events | From the start of the procedure up to 30 days post-procedure.
  The number and type of adverse events (AEs) and serious adverse events (SAEs), including but not limited to perforation, significant bleeding, and infection, are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, M.D., Ph.D., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided